CLINICAL TRIAL: NCT07055399
Title: Neoadjuvant Therapy of Iparomlimab and Tuvonralimab Combined With Chemotherapy-eclipse for Locally Advanced Cervical Cancer：A Single-arm, Open-label, Phase II Trial
Brief Title: Neoadjuvant Iparomlimab and Tuvonralimab Plus Chemotherapy-eclipse for Locally Advanced Cervical Cancer (NICE-CC)
Acronym: NICE-CC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Collaborators: Jiangsu Cancer Institute & Hospital (Other); Fuzhou University Affiliated Provincial Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NICE-CC trial
Record Dates: First submitted 2025-04-17; First posted 2025-07-08 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced Cervical Cancer
Keywords: Cervical Cancer; neoadjuvant; chemo-immunotherapy; iparomlimab and tuvonralimab;
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: The iparomlimab and tuvonralimab at a dosage of 5 mg/kg administered intravenously, along with cisplatin (75-80 mg/m², intravenously) and nab-paclitaxel (260 mg/m², intravenously) for one cycle. Then, two additional cycles (interval of 3 weeks) of iparomlimab and tuvonralimab (5 mg/kg, intravenously) were followed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group : iparomlimab and tuvonralimab plus nab-paclitaxel, cisplatin (Experimental): Participants will receive iparomlimab and tuvonralimab at a dose of 5 mg/kg, nab-paclitaxel at 260 mg/m², and cisplatin at 75-80 mg/m², all administered intravenously on day 1. After three weeks, participants will continue with only iparomlimab and tuvonralimab(5 mg/kg) for two additional cycles at an interval of 3 weeks.
  Interventions: Drug: neoadjuvant chemo-immunotherapy: Iparomlimab and tuvonralimab plus cisplatin,nab-paclitaxel for 1 cycle and Iparomlimab and tuvonralimab for 2 cycles

INTERVENTIONS:
Drug: neoadjuvant chemo-immunotherapy: Iparomlimab and tuvonralimab plus cisplatin,nab-paclitaxel for 1 cycle and Iparomlimab and tuvonralimab for 2 cycles — Neoadjuvant chemo-immunotherapy: Iparomlimab and tuvonralimab, cisplatin, and nab-paclitaxel for 1 cycle, then Iparomlimab and tuvonralimab continued for 2 cycles at 3-week intervals. Details:
  Iparomlimab and tuvonralimab 5 mg/kg, IV infusion, Q3W for 3 cycles Cisplatin：75-80 mg/m2, IV infusion, (cycle 1) Nab-paclitaxel 260 mg/m2，30min，IV infusion,(cycle 1)

SUMMARY:
Locally advanced cervical cancer (LACC) remains a significant global health concern with limited treatment options. Recent advancements suggest that using neoadjuvant anti-PD-1 inhibitors in combination with chemotherapy, followed by radical surgery, may be an effective treatment strategy for patients with PD-L1-positive LACC. This study aims to evaluate the efficacy and safety of preoperative treatment with iparomlimab and tuvonralimab-a bifunctional PD-1/CTLA-4 dual blocker-combined with chemotherapy for LACC.

DETAILED DESCRIPTION:
A total of 43 patients with FIGO 2018 stages IB3, IIA2, IIB, or IIIC1r will receive a combination treatment consisting of iparomlimab and tuvonralimab (5 mg/kg administered intravenously), cisplatin (75-80 mg/m², intravenously), and nab-paclitaxel (260 mg/m², intravenously) for one cycle. Following this, patients will receive two additional cycles of iparomlimab and tuvonralimab at the same dosage of 5 mg/kg, administered at three-week intervals. After completing three cycles of neoadjuvant treatment, patients who show a complete response (CR) or partial response (PR) will undergo radical surgery. The decision regarding subsequent adjuvant therapy will be guided by the NCCN guidelines. In contrast, patients with stable or progressive disease will proceed to concurrent chemoradiotherapy (CCRT).

ELIGIBILITY:
Inclusion Criteria:

* 1、Written informed consent
* 2、18-70 years old
* 3、Adequate organ function and ECOG of 0 ~1
* 4、Without systemic therapy at the time of enrollment
* 5、FIGO 2018 stage IB3, IIA2, or IIIC1r
* 6、Histologically confirmed squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the cervix
* 7、Measurable lesions could be defined by RECIST v1.1
* 8、Willing to get blood/ tumor tissue tested
* 9、Patients who observed the rules about the scheduled visit, study schedule, and medical examination
* 10、The function of major organs is normal, and the following criteria are met:
* 10.1 Blood routine examination must meet: (no blood transfusion within 14 days)

Hb≥90g/L:

ANC≥1.5x10^9/L; PLT≥100x10^9/L;

* 10.2 The biochemical examination must meet the following standards BIL < 1.5 × ULN; ALT and AST < 2.5xULN; ALB≥ 28 g/L
* 11、Patients who are willing and able to comply with visiting arrangements, treatment plans, laboratory tests, and other research procedures.

Exclusion Criteria:

* 1、History of other malignancies within 3 years
* 2、Participate in other clinical trials at the same time
* 3、Active autoimmune disease, which needs systemic therapy
* 4、Uncontrolled infection, which needs systemic therapy
* 5、History of allogeneic tissue/solid organ transplant
* 6、Serious illness, such as severe mental disorders, cardiac disease, coagulation disorders, digestive system disease, etc
* 7、Active HBV, HCV, or HIV infection
* 8、Pregnant or lactating female patients
* 9、Drug or alcohol abuse
* 10、 Unable or unwilling to sign the informed consent

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | From enrollment to the end of surgery at 3 months
  Pathological complete response（pCR） is defined as the absence of viable tumor cells by surgery

SECONDARY OUTCOMES:
Objective response rate (ORR) | From enrollment to the end of surgery at 3 months
  ORR is defined as the proportion of patients who achieve either a complete or partial response, as assessed by two experienced medical oncologists according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Event-free survival (EFS) | Through the study completion, an average of 2 year
  EFS is defined as the time from initial treatment to the date of disease progression that prevents definitive surgery, local or distant recurrence, occurrence of a second primary cancer, or death from any cause, whichever occurs first.
Primary pathological response (MPR) | From enrollment to the end of surgery at 3 months
  MPR is defined as having no more than 10% viable tumor by surgery.
Disease-free survival (DFS) | Through the study completion, an average of 2 year
  DFS is the interval from the initial treatment to the first occurrence of locoregional failure, distant metastasis, or death from any cause.
Adverse events | During the treatment（12months）
  Incidence of Treatment-Emergent Adverse Events, Including adverse events and complications. Incidence of adverse events using CTCAE 5.0; grade 3 treatment-related adverse events and higher-grade will be reported

OTHER OUTCOMES:
Immunophenotyping of peripheral blood mononuclear cells will be performed by flow cytometry | Samples taken prior/after to every cycle of treatment, or at progression, an average of 2 year
  Using flow cytometry to analyze the peripheral blood mononuclear cells to predict the efficacy of neoadjuvant chemo-immunotherapy. Results will be summarized by dose level
Tumor micrioenviroment assessment | Samples taken prior/after to every cycle of treatment, or at progression, an average of 2 year
  using tumor tissue (multiple immunofluorescence) to assess immune cells before and after 3 cycles of neoadjuvant chemo-immunotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No
Not yet decided

REFERENCES:
- [Background] Wu X, Sun Y, Yang H, Wang J, Lou H, Li D, Wang K, Zhang H, Wu T, Li Y, Wang C, Li G, Wang Y, Li D, Tang Y, Pan M, Cai H, Wang W, Yang B, Qian H, Tian Q, Yao D, Cheng Y, Wei B, Li X, Wang T, Hao M, Wang X, Wang T, Ran J, Zhu H, Zhu L, Liu X, Li Y, Chen L, Li Q, Yan X, Wang F, Cai H, Zhang Y, Liang Z, Liu F, Huang Y, Xia B, Qu P, Zhu G, Chen Y, Song K, Sun M, Chen Z, Zhou Q, Hu L, Abulizi G, Guo H, Liao S, Ye Y, Yan P, Tang Q, Sun G, Liu T, Lu D, Hu M, Wang ZM, Li B, Xia M. Cadonilimab plus platinum-based chemotherapy with or without bevacizumab as first-line treatment for persistent, recurrent, or metastatic cervical cancer (COMPASSION-16): a randomised, double-blind, placebo-controlled phase 3 trial in China. Lancet. 2024 Oct 26;404(10463):1668-1676. doi: 10.1016/S0140-6736(24)02135-4. Epub 2024 Oct 16. PMID 39426385
- [Background] Nederlof I, Isaeva OI, de Graaf M, Gielen RCAM, Bakker NAM, Rolfes AL, Garner H, Boeckx B, Traets JJH, Mandjes IAM, de Maaker M, van Brussel T, Chelushkin M, Champanhet E, Lopez-Yurda M, van de Vijver K, van den Berg JG, Hofland I, Klioueva N, Mann RM, Loo CE, van Duijnhoven FH, Skinner V, Luykx S, Kerver E, Kalashnikova E, van Dongen MGJ, Sonke GS, Linn SC, Blank CU, de Visser KE, Salgado R, Wessels LFA, Drukker CA, Schumacher TN, Horlings HM, Lambrechts D, Kok M. Neoadjuvant nivolumab or nivolumab plus ipilimumab in early-stage triple-negative breast cancer: a phase 2 adaptive trial. Nat Med. 2024 Nov;30(11):3223-3235. doi: 10.1038/s41591-024-03249-3. Epub 2024 Sep 16. PMID 39284953
- [Background] Keam SJ. Iparomlimab and Tuvonralimab: First Approval. Drugs. 2025 May;85(5):699-706. doi: 10.1007/s40265-025-02160-6. Epub 2025 Apr 1. PMID 40167968
- [Background] Li K, Chen J, Hu Y, Wang YZ, Shen Y, Chen G, Peng W, Fang Z, Xia B, Chen X, Song K, Wang Y, Zou D, Wang YC, Han Y, Feng X, Yuan J, Guo S, Meng X, Feng C, Chen Y, Yang J, Fan J, Wang J, Ai J, Ma D, Sun C. Neoadjuvant chemotherapy plus camrelizumab for locally advanced cervical cancer (NACI study): a multicentre, single-arm, phase 2 trial. Lancet Oncol. 2024 Jan;25(1):76-85. doi: 10.1016/S1470-2045(23)00531-4. Epub 2023 Dec 1. PMID 38048802
- [Background] Miriyala R, Mahantshetty U, Maheshwari A, Gupta S. Neoadjuvant chemotherapy followed by surgery in cervical cancer: past, present and future. Int J Gynecol Cancer. 2022 Mar;32(3):260-265. doi: 10.1136/ijgc-2021-002531. PMID 35256411
- [Background] Abu-Rustum NR, Yashar CM, Arend R, Barber E, Bradley K, Brooks R, Campos SM, Chino J, Chon HS, Crispens MA, Damast S, Fisher CM, Frederick P, Gaffney DK, Gaillard S, Giuntoli R, Glaser S, Holmes J, Howitt BE, Lea J, Mantia-Smaldone G, Mariani A, Mutch D, Nagel C, Nekhlyudov L, Podoll M, Rodabaugh K, Salani R, Schorge J, Siedel J, Sisodia R, Soliman P, Ueda S, Urban R, Wyse E, McMillian NR, Aggarwal S, Espinosa S. NCCN Guidelines(R) Insights: Cervical Cancer, Version 1.2024. J Natl Compr Canc Netw. 2023 Dec;21(12):1224-1233. doi: 10.6004/jnccn.2023.0062. PMID 38081139
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751